CLINICAL TRIAL: NCT02984111
Title: Placebo- Controlled,Randomized,Double Blind Trial of Erythropoietin Effect on Ischemic_ Reperfusion Injury in Coronary Artery Bypass Graft Surgery
Brief Title: Erythropoietin Effect on Ischemic_ Reperfusion Injury in Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Collaborators: Pooyesh Darou (Other)
Responsible Party: Principal Investigator, Mahnoosh Foroughi, Clinical Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IR.sbmu.ram.rec.1394.292; IRCT2016011621087N1 (Registry Identifier: Iranian registry of clinical trial)
Record Dates: First submitted 2016-11-13; First posted 2016-12-06 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Myocardial Ischemic Reperfusion Injury
Keywords: Coronary artery bypass; Erythropoietin; Inflammation; IL-6; Reperfusion injury; YKL- 40
MeSH Terms: conditions — Myocardial Reperfusion Injury; Inflammation; Reperfusion Injury | interventions — Saline Solution; Erythropoietin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- group A (Active Comparator): 20000 IU erythropoietin infusion during aortic cross clamp in 45-60 minutes
  Interventions: Drug: erythropoietin
- group B (Active Comparator): 20000 IU erythropoietin infusion after induction of anesthesia and before undergoing cardiopulmonary bypass pump in 45-60 minutes
  Interventions: Drug: erythropoietin
- control (Placebo Comparator): 50 ml normal saline infusion during aortic cross clamp in 45-60 minutes
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: normal saline
  Other Names: N/S
  Arms: control
Drug: erythropoietin
  Other Names: epoietin alfa
  Arms: group A; group B

SUMMARY:
The aim of this trail is to assess the safety and therapeutic effects of single EPO intervention in different times during coronary surgery in changes of inflammatory response.

DETAILED DESCRIPTION:
In addition to well-known effect of Erythropoietin (EPO) on erythropoiesis in hypoxic conditions, some lines of evidence suggest its protective effects against reperfusion injury in several tissues by its specific receptor.

Preclinical studies have indicated a broad variety of cardioprotective actions for EPO. It improves cardiac function and exercise capacity in congestive heart failure, angiogenesis, limit myocardial inflammatory response, cardiac remodeling, infarct size and apoptosis extension induced by reperfusion injury. Activation of EPO receptor in endothelial and cardiac cells is suggested to attenuate proinflammatory cytokines production and inflammatory cells infiltration, and increasing nitric oxide production through possible mechanisms.

Reperfusion injury is unavoidable event during cardiac surgery using cardiopulmonary bypass.It is associated with inflammation, cell injury and attenuate contractility property.

Although it is an area of concern and many clinical studies have been designed by different interventions, it remains a major challenge. EPO intervention during heart reperfusion (surgery/ percutaneous angioplasty) as a new promise of cardioprotection strategy is the main design of several studies with conflicting results .

ELIGIBILITY:
Inclusion Criteria:

* Revascularization requirement according to angiographic evidence
* Elective coronary artery bypass graft surgery
* First time coronary artery bypass graft surgery
* On-pump coronary artery bypass graft surgery

Exclusion Criteria:

* History of myocardial infarction in the past 3 months
* Previous myocardial trauma or major surgery in the past 3 months
* Cr>2mg/dl
* Receiving streptokinase or previous reperfusion treatments
* Erythropoietin intake in the recent 6 months
* Known thromboembolic disorder and malignant disease
* Uncontrolled hypertension
* Polycythemia
* Previous valvular surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in Interleukin 6(IL6) | Change from baseline until 48 hours after surgery
  Serum IL6(an inflammatory marker) level is measured before operation (base),just after operation,24 hours after operation,48 hours after operation
Change in YKL-40 | Change from baseline until 48 hours after surgery
  Chitinase-3-like protein 1 (CHI3L1), also known as YKL-40 is an inflammatory marker.Serum YKL-40 level is measured before operation (base),just after operation,24 hours after operation,48 hours after operation
Change in pro b-type natriuretic peptide(pro BNP) | Change from baseline until 48 hours after surgery
  Serum pro BNP level is measured before operation (base),just after operation,24 hours after operation,48 hours after operation

SECONDARY OUTCOMES:
Volume of bleeding | During operation until 24 hours after surgery
Need to blood transfusion | During and after operation, through study completion,an average of one week
  Number of packed cell and fresh frozen plasma that transfused in the period of time that patient is hospitalized.
Ventilation time | Period of time after surgery that patient has been intubated in ICU,an average of 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mahnoosh Foroughi, MD,, Principal Investigator — Cardiovascular Research Center, Shahid Beheshti University of Medical Sciences. Tehran, Iran.
Locations (1):
- Cardiovascular Research Center, Shahid Beheshti University of Medical Sciences., Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziabakhsh-Tabary S, Jalalian R, Mokhtari-Esbuie F, Habibi MR. Echocardiographic Evaluation of the Effects of a Single Bolus of Erythropoietin on Reducing Ischemia-Reperfusion Injuries during Coronary Artery Bypass Graft Surgery; A Randomized, Double-Blind, Placebo-Control Study. Iran J Med Sci. 2014 Mar;39(2):94-101. PMID 24644377
- [Background] Ludman AJ, Yellon DM, Hasleton J, Ariti C, Babu GG, Boston-Griffiths E, Venugopal V, Walker M, Holdright D, Swanton H, Crake T, Brull D, Moon JC, Puranik R, Muthurangu V, Taylor A, Hausenloy DJ. Effect of erythropoietin as an adjunct to primary percutaneous coronary intervention: a randomised controlled clinical trial. Heart. 2011 Oct;97(19):1560-5. doi: 10.1136/hrt.2011.223867. PMID 21900585
- [Background] Joyeux-Faure M, Durand M, Bedague D, Protar D, Incagnoli P, Paris A, Ribuot C, Levy P, Chavanon O. Evaluation of the effect of one large dose of erythropoietin against cardiac and cerebral ischemic injury occurring during cardiac surgery with cardiopulmonary bypass: a randomized double-blind placebo-controlled pilot study. Fundam Clin Pharmacol. 2012 Dec;26(6):761-70. doi: 10.1111/j.1472-8206.2011.00992.x. Epub 2011 Sep 20. PMID 21929528
- [Background] Najjar SS, Rao SV, Melloni C, Raman SV, Povsic TJ, Melton L, Barsness GW, Prather K, Heitner JF, Kilaru R, Gruberg L, Hasselblad V, Greenbaum AB, Patel M, Kim RJ, Talan M, Ferrucci L, Longo DL, Lakatta EG, Harrington RA; REVEAL Investigators. Intravenous erythropoietin in patients with ST-segment elevation myocardial infarction: REVEAL: a randomized controlled trial. JAMA. 2011 May 11;305(18):1863-72. doi: 10.1001/jama.2011.592. PMID 21558517
- [Background] Ott I, Schulz S, Mehilli J, Fichtner S, Hadamitzky M, Hoppe K, Ibrahim T, Martinoff S, Massberg S, Laugwitz KL, Dirschinger J, Schwaiger M, Kastrati A, Schmig A; REVIVAL-3 Study Investigators. Erythropoietin in patients with acute ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention: a randomized, double-blind trial. Circ Cardiovasc Interv. 2010 Oct;3(5):408-13. doi: 10.1161/CIRCINTERVENTIONS.109.904425. Epub 2010 Aug 24. PMID 20736448
- [Result] Vilarinho KA, de Oliveira PP, Saad MJ, Eghtesady P, Filho LM, Vieira RW, Petrucci O. Erythropoietin protects the systolic function of neonatal hearts against ischaemia/reperfusion injury. Eur J Cardiothorac Surg. 2013 Jan;43(1):156-62. doi: 10.1093/ejcts/ezs254. Epub 2012 May 7. PMID 22564802
- [Result] Watson AJ, Gao L, Sun L, Tsun J, Jabbour A, Ru Qiu M, Jansz PC, Hicks M, Macdonald PS. Enhanced preservation of the rat heart after prolonged hypothermic ischemia with erythropoietin-supplemented Celsior solution. J Heart Lung Transplant. 2013 Jun;32(6):633-40. doi: 10.1016/j.healun.2013.03.014. PMID 23701853
- [Result] Lu MJ, Chen YS, Huang HS, Ma MC. Erythropoietin alleviates post-ischemic injury of rat hearts by attenuating nitrosative stress. Life Sci. 2012 May 22;90(19-20):776-84. doi: 10.1016/j.lfs.2012.04.012. Epub 2012 Apr 12. PMID 22521289
- [Result] Xu X, Cao Z, Cao B, Li J, Guo L, Que L, Ha T, Chen Q, Li C, Li Y. Carbamylated erythropoietin protects the myocardium from acute ischemia/reperfusion injury through a PI3K/Akt-dependent mechanism. Surgery. 2009 Sep;146(3):506-14. doi: 10.1016/j.surg.2009.03.022. Epub 2009 Jun 9. PMID 19715808
- [Result] Prunier F, Biere L, Gilard M, Boschat J, Mouquet F, Bauchart JJ, Charbonnier B, Genee O, Guerin P, Warin-Fresse K, Durand E, Lafont A, Christiaens L, Abi-Khalil W, Delepine S, Benard T, Furber A. Single high-dose erythropoietin administration immediately after reperfusion in patients with ST-segment elevation myocardial infarction: results of the erythropoietin in myocardial infarction trial. Am Heart J. 2012 Feb;163(2):200-7.e1. doi: 10.1016/j.ahj.2011.11.005. PMID 22305837
- [Result] Voors AA, Belonje AM, Zijlstra F, Hillege HL, Anker SD, Slart RH, Tio RA, van 't Hof A, Jukema JW, Peels HO, Henriques JP, Ten Berg JM, Vos J, van Gilst WH, van Veldhuisen DJ; HEBE III Investigators. A single dose of erythropoietin in ST-elevation myocardial infarction. Eur Heart J. 2010 Nov;31(21):2593-600. doi: 10.1093/eurheartj/ehq304. Epub 2010 Aug 29. PMID 20802250
- [Result] Momeni M, Liistro G, Baele P, Matta A, Kahn D, Van Dyck M, De Kock M, De Kerchove L, Glineur D, Thiry D, Gregoire A, Jacquet LM, Laarbui F, Watremez C. An increase in endogenous erythropoietin concentrations has no cardioprotective effects in patients undergoing coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2012 Apr;26(2):251-7. doi: 10.1053/j.jvca.2011.07.034. Epub 2011 Oct 5. PMID 21975293
- [Result] Taniguchi N, Nakamura T, Sawada T, Matsubara K, Furukawa K, Hadase M, Nakahara Y, Nakamura T, Matsubara H. Erythropoietin prevention trial of coronary restenosis and cardiac remodeling after ST-elevated acute myocardial infarction (EPOC-AMI): a pilot, randomized, placebo-controlled study. Circ J. 2010 Nov;74(11):2365-71. doi: 10.1253/circj.cj-10-0267. Epub 2010 Sep 8. PMID 20834185
- [Result] Bergmann MW, Haufe S, von Knobelsdorff-Brenkenhoff F, Mehling H, Wassmuth R, Munch I, Busjahn A, Schulz-Menger J, Jordan J, Luft FC, Dietz R. A pilot study of chronic, low-dose epoetin-beta following percutaneous coronary intervention suggests safety, feasibility, and efficacy in patients with symptomatic ischaemic heart failure. Eur J Heart Fail. 2011 May;13(5):560-8. doi: 10.1093/eurjhf/hfr002. PMID 21505058
- [Result] Ferrario M, Arbustini E, Massa M, Rosti V, Marziliano N, Raineri C, Campanelli R, Bertoletti A, De Ferrari GM, Klersy C, Angoli L, Bramucci E, Marinoni B, Ferlini M, Moretti E, Raisaro A, Repetto A, Schwartz PJ, Tavazzi L. High-dose erythropoietin in patients with acute myocardial infarction: a pilot, randomised, placebo-controlled study. Int J Cardiol. 2011 Feb 17;147(1):124-31. doi: 10.1016/j.ijcard.2009.10.028. Epub 2009 Nov 10. PMID 19906454
- [Result] Poulsen TD, Andersen LW, Steinbruchel D, Gotze JP, Jorgensen OS, Olsen NV. Two large preoperative doses of erythropoietin do not reduce the systemic inflammatory response to cardiac surgery. J Cardiothorac Vasc Anesth. 2009 Jun;23(3):316-23. doi: 10.1053/j.jvca.2008.08.018. Epub 2008 Oct 22. PMID 18948032
- [Result] Kagaya Y, Asaumi Y, Wang W, Takeda M, Nakano M, Satoh K, Fukumoto Y, Shimokawa H. Current perspectives on protective roles of erythropoietin in cardiovascular system: erythropoietin receptor as a novel therapeutic target. Tohoku J Exp Med. 2012 Jun;227(2):83-91. doi: 10.1620/tjem.227.83. PMID 22688525
- [Result] Gobe GC, Morais C, Vesey DA, Johnson DW. Use of high-dose erythropoietin for repair after injury: A comparison of outcomes in heart and kidney. J Nephropathol. 2013 Jul;2(3):154-65. doi: 10.12860/JNP.2013.27. Epub 2013 Jul 1. PMID 24475445